CLINICAL TRIAL: NCT00130481
Title: Pediatric Atorvastatin in Diabetes Intervention Trial (PADIT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 576-2004; GCRC M-01 RR 000082; Pfizer 2004-0926; DARE 187
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: Diabetes; Children; Adolescents; Arterial Compliance; Physiology Cardiovascular Endothelium
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin 20 mg daily for 3 months

SUMMARY:
The purpose of this study is to determine if Atorvastatin can improve blood vessel stiffness and blood vessel function in children 10-18 years old with Type 1 and Type 2 diabetes. Subjects will receive atorvastatin 20mg or placebo daily for 3 months and will then switch therapies for the next 3 months.

Hypothesis: Atorvastatin will improve blood vessel function by decreasing arterial stiffness and improving blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus (T1DM) or Type 2 Diabetes Mellitus (T2DM) for more than 1 year
* Age 10-18 years.

Exclusion Criteria:

* Cardiovascular disease (CVD)
* Liver disease
* Pregnancy
* Use of cholesterol or triglyceride lowering drugs
* Perceived inability to comply with the study protocol
* Endocrinopathy other than diabetes

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100
Dates: Start 2005-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Augmentation Index (arterial stiffness)
ENDO-PAT (Peripheral Arterial Tone) score (endothelial function)
Low density lipoprotein

SECONDARY OUTCOMES:
Urine microalbumin
Pubertal stage
Body mass index (BMI)
Blood pressure
Glycated hemoglobin (HbA1c)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Haller, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Haller MJ, Samyn M, Nichols WW, Brusko T, Wasserfall C, Schwartz RF, Atkinson M, Shuster JJ, Pierce GL, Silverstein JH. Radial artery tonometry demonstrates arterial stiffness in children with type 1 diabetes. Diabetes Care. 2004 Dec;27(12):2911-7. doi: 10.2337/diacare.27.12.2911. PMID 15562206
- [Derived] Haller MJ, Stein JM, Shuster JJ, Theriaque D, Samyn MM, Pepine C, Silverstein JH. Pediatric Atorvastatin in Diabetes Trial (PADIT): a pilot study to determine the effect of atorvastatin on arterial stiffness and endothelial function in children with type 1 diabetes mellitus. J Pediatr Endocrinol Metab. 2009 Jan;22(1):65-8. doi: 10.1515/jpem.2009.22.1.65. PMID 19344076